CLINICAL TRIAL: NCT00364195
Title: A Pharmacokinetic Interaction and Safety and Efficacy Phase II, Open Label Study With a Safety Lead-in Evaluating Docetaxel Plus Tesmilifene (YMB1002) in Patients With Metastatic Breast Cancer Suitable for Treatment With Docetaxel
Brief Title: Tesmilifene in Combination With Docetaxel in the Treatment of Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: YM BioSciences (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YMB1002 203
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer; Tesmilifene; DPPE
MeSH Terms: conditions — Breast Neoplasms | interventions — tesmilifene

INTERVENTIONS:
Drug: Tesmilifene (YMB1002)

SUMMARY:
This is a Phase II study designed to evaluate whether the co-administration of a fixed dose of tesmilifene and a standard regimen of docetaxel alters the plasma pharmacokinetics of docetaxel. This study will also assess the safety and efficacy of the tesmilifene/docetaxel combination in metastatic breast cancer patients.

DETAILED DESCRIPTION:
Primary Objective:

1. To evaluate whether the co-administration of a fixed dose of tesmilifene (5.3 mg/kg) with a standard dose of docetaxel (100 mg/m2) alters the plasma pharmacokinetics of docetaxel compared to the pharmacokinetics of docetaxel when given alone.

Secondary Objectives:

1. To correlate plasma tesmilifene levels during and following the infusion with the acute tesmilifene-related adverse events observed during and after the infusion.
2. To collect safety information for tesmilifene when administered in combination with docetaxel.
3. To evaluate response rate, duration of response and overall survival in metastatic breast cancer patients receiving docetaxel plus tesmilifene.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with documented histological/cytological proof of metastatic and/or recurrent breast cancer suitable for treatment with docetaxel
2. Patients must have documented hormone receptor status (ER/PR) and Her-2 neu status determined either by Immunohistochemistry or FISH, within 21 days of randomisation, if possible, otherwise receptor status from patient history can be used, if determined from earlier biopsy/surgery. Patients may be randomised whilst results of hormone receptor status (ER/PR) and Her-2 neu status are pending from the laboratory.
3. Radiological investigations must be conducted within 21 days prior to randomization. Exceptions will be made only for patients who have had NEGATIVE examinations with 35 days prior to randomisation.
4. Presence of at least one uni-dimensional measurable lesion. 5. Disease free interval (DFI) less than or equal to 24 months (from the time of initial surgery to randomization date).

6. Previous hormone therapy, chemotherapy and radiation therapy allowed as defined in the protocol 7. Patients with an ECOG status of 0, 1 or 2. 8. Have a life expectancy of at least 6 months 9. Patients must be female and aged ≥ 18 years and ≤ 65 years 10. Patients must be willing and able to follow instructions and make all required study visits.

11. Patients must be willing and able to give written consent to participate in this study.

12. Patients must have adequate organ and marrow function as defined in the protocol.

13. All women of child-bearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity of 25 IU/L of BHCG) within 72 hours prior to randomization.

14. Patients must have a negative blood tests for HIV and Hepatitis B and C within 4 weeks prior to randomisation.

Exclusion Criteria:

1. Patients with previous malignancies, excluding curatively treated basal or squamous cell carcinoma of the skin or in-situ cervical cancer or any other cancer treated more than five years prior to study entry and presumed cured.
2. Patients with known brain or meningeal metastases (CT scan not required to rule this out unless there is a clinical suspicion of CNS disease).
3. Patients whose only measurable disease is in the bone.
4. Patients using chemotherapeutic agents for any malignancy within 4 weeks prior to study entry or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
5. Patients who have received treatment with any other investigational drug within the preceding 4 weeks.
6. Patient who have received hormone treatment for cancer within 6 weeks or 5 half-lives of enrolment (whichever is shorter).
7. Pregnant and breast-feeding females.
8. Patients with history of seizure disorder.
9. Patients with clinically significant cardiovascular, pulmonary, renal, endocrine, hepatic, respiratory, neurologic, psychiatric, immunologic, gastrointestinal, haematologic, metabolic or any other condition or laboratory abnormality that, in the opinion of the Investigator or Medical Director of YM BioSciences Inc., makes the patient unsuitable for participation in the study.
10. Known allergy or hypersensitivity to test article ingredients.
11. Patients on COX 1 or 2 prostaglandin inhibitors (e.g. ASA, other NSAID's, Celebrex®, Vioxx® ) who can not comply with guidelines or concomitant therapy as outlined in appendix V, i.e.; avoid from midnight before treatment until midnight post treatment. Patients who are required to take low dose aspirin (81 mg) may be allowed to continue taking low dose aspirin.
12. Patients on H1 antagonists (e.g., antihistamines, antidepressants or antiemetics) detailed in appendix V who can not comply with guidelines or concomitant therapy as outlined in appendix V, i.e.; avoid from 12 hours before the start of protocol treatment begins until the patient is off protocol treatment.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2006-06

PRIMARY OUTCOMES:
To evaluate whether the co-administration of a fixed dose of tesmilifene (5.3 mg/kg) with a standard dose of docetaxel (100 mg/m2) alters the plasma pharmacokinetics of docetaxel compared to the pharmacokinetics of docetaxel when given alone.

SECONDARY OUTCOMES:
To correlate plasma tesmilifene levels during and following the infusion with the acute tesmilifene-related adverse events observed during and after the infusion.
To collect safety information for tesmilifene when administered in combination with docetaxel.
To evaluate response rate, duration of response and overall survival in metastatic breast cancer patients receiving docetaxel plus tesmilifene.

CONTACTS AND LOCATIONS:
Locations (3):
- Serbia (3):
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Institute for Oncology and Radiology of Serbia (IORS), Belgrade
  - Institute of Oncology Sremska Kamenica, Kamenitz